CLINICAL TRIAL: NCT06088849
Title: Maternal Treatment With ACE-inhibitors and Breastfeeding: a Mono-centric Study on the Exposure Through Breast Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S65657
Record Dates: First submitted 2022-05-06; First posted 2023-10-18 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Breast Feeding; Hypertension; Heart Failure; Proteinuria
Keywords: Angiotensin-converting-enzyme inhibitor
MeSH Terms: conditions — Breast Feeding; Hypertension; Heart Failure; Proteinuria | interventions — Phlebotomy

STUDY DESIGN:
Intervention Model Description: We will enroll mothers who have been prescribed ACE-inhibitors for medical reasons and are breastfeeding their infant while taking this medication. The mother will be asked to collect milk samples and donate 2 blood samples during a 24h period. Furthermore, we will ask the parents if we can collect a blood sample of the child. In addition, clinical maternal and infant variables will be collected, as well as medication intake, sampling information and general infant health.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lactating mothers taking ACE-inhibitors (Other): Lactating mothers who are breastfeeding their infant (0-6 months) while taking ACE-inhibitors.
  Interventions: Procedure: Venipuncture

INTERVENTIONS:
Procedure: Venipuncture — The lactating mother will be asked to collect milk samples and donate 2 blood samples, which is not a part of their normal follow-up/treatment. We will also aks the parents if we can collect a blood sample fo the infant (0-6 months).
  Other Names: Venipuncture infant

SUMMARY:
The ACE-inhibitors is one group of essential medication for which reliable data on the safety during breastfeeding is lacking. ACE inhibitors are indicated for several severe or life-threatening disorders like hypertension, heart failure or nephrotic range proteinuria and diabetic nephropathy. However, data on the transfer of ACE inhibitors into the human breast milk remains very limited. After delivery, ACE inhibitor therapy is often postponed if the mother is breastfeeding, requiring multiple other medications to control the disease, or switched from long to short acting forms, decreasing therapeutic adherence. Limited available data shows that the transfer of ACE-inhibitors into the milk is probably low, and thus that ACE-inhibitor are likely to be safe during breastfeeding.

The objective of this trial is to collect information about the breast milk transfer, and subsequent infant exposure and general health outcome to selected maternal medication (ACE inhibitors) in patients from UZ Leuven. Furthermore, we will also use these data to verify the predictive performance of physiologically-based pharmacokinetic models to predict breast milk and subsequent neonatal exposure to maternal medication during lactation. The medicines that will be investigated are perindopril, captopril, cilazapril, enalapril, fosinopril, lisinopril, quinapril, ramipril and zofenopril.

The investigators will enroll +/-10 mothers, who have been prescribed ACE inhibitors for medical reasons and are breastfeeding their infant while taking this medication.The mother will be asked to collect milk samples during 24 h and 2 blood samples: one at the time of milk pumping the first time after medication intake, and one at the last pumping session of the 24 h. Furthermore, we will ask the parents if we can collect a blood sample of the child (1mL/kg, and max 2,5mL). In addition, clinical maternal and infant variables will be collected, as well as medication intake, sampling information and general infant health.

To conclude, with this study we hope to generate human data about the use of ACE inhibitors during breastfeeding. This information is an essential first step towards evidence-based risk assessment on the use of these drugs during lactation.

ELIGIBILITY:
Inclusion Criteria:

For lactating mothers

* Lactating
* 0-6 months postpartum
* Age: ≥18 year
* On steady state ACE-inhibitor therapy, for any indication (e.g. perindopril, captopril, cilazapril, enalapril, fosinopril, lisinopril, quinapril, ramipril & zofenopril)
* Willing to express breast milk
* Informed consent to participate and for processing their personal data

For neonates/infants

* 0-6 months of age at inclusion of the mother
* Postmenstrual age: ≥ 37 weeks
* In case of blood sampling: exclusively breastfed at the time of sampling
* Parental informed consent to participate and for processing their personal data

Exclusion Criteria:

* Participation in a trial with an investigational product within the previous three months
* Not meeting the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The secretion rates of ACE-inhibitors into the human breast milk | 24 hours (sampling day)
  The maternal plasma concentration, milk-to-plasma ratios fo the selected medicines, PK parameters of the parent medication and metabolites in mature breast milk, such as area under the milk concentration-time curve (AUC), the average concentration, peak and trough milk concentrations and time to reach peak milk concentration.

SECONDARY OUTCOMES:
The child's systemic exposure after exposure to ACE-inhibitors via breastfeeding | during the sampling day (24 hours)
  The infant's plasma concentration of ACE-inhibitors (if a blood sample of the infant is obtained), the relevant infant dose, the daily infant dose, the infant/maternal plasma ratio (if a blood sample of the neonate is obtained) after exposure to maternal ACE-inhibitors via breastfeeding.
The child's outcome after exposure to ACE-inhibitors via breastfeeding | Up to 2 months after inclusion
  The health condition of the infants after exposure to maternal ACE-inhibitors via breastfeeding.

CONTACTS AND LOCATIONS:
Overall Officials: Kristel Van Calsteren, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson PO. Drugs in Lactation. Pharm Res. 2018 Feb 6;35(3):45. doi: 10.1007/s11095-017-2287-z. PMID 29411152
- [Background] Koshimichi H, Ito K, Hisaka A, Honma M, Suzuki H. Analysis and prediction of drug transfer into human milk taking into consideration secretion and reuptake clearances across the mammary epithelia. Drug Metab Dispos. 2011 Dec;39(12):2370-80. doi: 10.1124/dmd.111.040972. Epub 2011 Sep 22. PMID 21940904
- [Background] Ito N, Ito K, Ikebuchi Y, Toyoda Y, Takada T, Hisaka A, Oka A, Suzuki H. Prediction of Drug Transfer into Milk Considering Breast Cancer Resistance Protein (BCRP)-Mediated Transport. Pharm Res. 2015 Aug;32(8):2527-37. doi: 10.1007/s11095-015-1641-2. Epub 2015 Feb 19. PMID 25690342
- [Background] McNamara PJ, Burgio D, Yoo SD. Pharmacokinetics of cimetidine during lactation: species differences in cimetidine transport into rat and rabbit milk. J Pharmacol Exp Ther. 1992 Jun;261(3):918-23. PMID 1602396
- [Background] Kimura S, Morimoto K, Okamoto H, Ueda H, Kobayashi D, Kobayashi J, Morimoto Y. Development of a human mammary epithelial cell culture model for evaluation of drug transfer into milk. Arch Pharm Res. 2006 May;29(5):424-9. doi: 10.1007/BF02968594. PMID 16756089
- [Background] Garessus EDG, Mielke H, Gundert-Remy U. Exposure of Infants to Isoniazid via Breast Milk After Maternal Drug Intake of Recommended Doses Is Clinically Insignificant Irrespective of Metaboliser Status. A Physiologically-Based Pharmacokinetic (PBPK) Modelling Approach to Estimate Drug Exposure of Infants via Breast-Feeding. Front Pharmacol. 2019 Jan 22;10:5. doi: 10.3389/fphar.2019.00005. eCollection 2019. PMID 30723406
- [Background] Piepho RW. Overview of the angiotensin-converting-enzyme inhibitors. Am J Health Syst Pharm. 2000 Oct 1;57 Suppl 1:S3-7. doi: 10.1093/ajhp/57.suppl_1.S3. PMID 11030016
- [Background] Jones HM, Mayawala K, Poulin P. Dose selection based on physiologically based pharmacokinetic (PBPK) approaches. AAPS J. 2013 Apr;15(2):377-87. doi: 10.1208/s12248-012-9446-2. Epub 2012 Dec 27. PMID 23269526
- [Background] Mould DR, Upton RN. Basic concepts in population modeling, simulation, and model-based drug development-part 2: introduction to pharmacokinetic modeling methods. CPT Pharmacometrics Syst Pharmacol. 2013 Apr 17;2(4):e38. doi: 10.1038/psp.2013.14. No abstract available. PMID 23887688
- [Background] FDA. Clinical Lactation Studies: Considerations for Study Design Guidance for Industry DRAFT GUIDANCE. May 2019.
- See also: Breastfeeding — https://www.who.int/health-topics/breastfeeding#tab=tab_1